CLINICAL TRIAL: NCT02216825
Title: Effect of L. Reuteri NCIMB 30242 on Plasma Bile Acid Profile
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Micropharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: MP-12LCHMe
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-06

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed release capsule, L. reuteri NCIMB 30242 (Experimental)
  Interventions: Dietary Supplement: Delayed release capsule, L. reuteri NCIMB 30242, escalated dose
- Standard vegetarian capsule, L. reuteri NCIMB 30242 (Experimental)
  Interventions: Dietary Supplement: Standard vegetarian capsule, L. reuteri NCIMB 30242, escalated dose

INTERVENTIONS:
Dietary Supplement: Delayed release capsule, L. reuteri NCIMB 30242, escalated dose
  Arms: Delayed release capsule, L. reuteri NCIMB 30242
Dietary Supplement: Standard vegetarian capsule, L. reuteri NCIMB 30242, escalated dose
  Arms: Standard vegetarian capsule, L. reuteri NCIMB 30242

SUMMARY:
Background: In recent years, probiotics have shown promise in treating a variety of diseases. Previously, the investigators have reported on the clinical efficacy of bile salt hydrolase active Lactobacillus reuteri NCIMB 30242 in improving the lipid profile in hypercholesterolemic adults.

Objective: The purpose of the study is to investigate the effect of a delayed release or standard vegetarian capsule containing L. reuteri NCIMB 30242, taken in escalated dose over a 4 week period, on the plasma bile acid profile.

Design: The study design is a pilot, randomized, double-blind, dose-escalation study. The study will last a total of 6 weeks, including a 4-week intervention period and a 2-week washout period.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, aged 20 to 75 years (bounds included).
* LDL-C ≥ 3.40 mmol/L.
* TG < 4.00 mmol/L.
* TBA < 10 umol/L.
* BMI range from 23.0 to 32.5 kg/m2 (bounds included).
* Signed informed consent form prior to inclusion in the study.
* Note: Subjects will be permitted to take stable doses of thyroid hormone and anti-hypertensive agents, as long as these are continued equivalently throughout the duration of study.
* Female subjects not of child bearing potential. Defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation) OR Female subject of childbearing potential who agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include: Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System); Intrauterine devices; Vasectomy of partner; Total abstinence.

Exclusion Criteria:

* Use of cholesterol lowering prescription drugs within the last 6 months.
* Use of plant sterols, omega 3, fish oil, soy protein, soluble oat fiber, psyllium seed husk, or other cholesterol lowering non-prescription supplements within last 1 month.
* History of chronic use of alcohol (> 2 drinks/d).
* History of heavy smoking (≥ 20 cigarettes/d).
* Use of systemic antibodies, corticosteroids, androgens, or phenytoin.
* Immune-compromised subjects (e.g. AIDS, lymphoma, subjects undergoing long-term corticosteroid treatment)
* Subject having experienced any cardiovascular event (Myocardial infarction, coronary artery bypass, or other major surgical procedures) in the last 6 months.
* Subjects with elevated LDL-C (≥ 3.40 mmol/L) and high (>20%) CVD risk estimated by the Framingham risk score
* Previously diagnosed Type I or Type II diabetes.
* Subject receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters.
* Subject currently involved in a clinical trial or in an exclusion period following participation in another clinical trial.
* History of angina, congestive heart failure, inflammatory bowel disease, pancreatitis, gastrointestinal, renal, pulmonary, hepatic or biliary disease, or cancer (evidence of active lesions, chemotherapy or surgery in the past year).
* Clinically significant abnormal laboratory results at screening.
* Chronic user of probiotics or fibre laxative (greater than 2 doses/wk), or stimulant laxatives.
* History of eating disorders.
* Exercise greater than 15 miles/wk or 4,000 kcal/wk.
* Female subjects that are pregnant, breast feeding or intend to get pregnant.
* Allergy or sensitivity to test product ingredients
* Allergy or sensitivity to all 3 antibiotics (Clindamycin, Erythromycin and Ampicillin).

Ages: 20 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the change in plasma bile acid profile from baseline to endpoint | Week 0 and Week 4 of intervention period